CLINICAL TRIAL: NCT04304456
Title: Epidemiology and Determinants of Outcomes of Hospital Acquired Blood Stream Infections in the Intensive Care in Turkey
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: SCARE (Study group for carbapenem resistance) (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: KA-19126
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Bacteremia; Sepsis; Hospital Acquired Condition
Keywords: Bacteremia; Antimicrobial resistance; Mortality; Hospital acquired infections
MeSH Terms: conditions — Bacteremia; Sepsis; Iatrogenic Disease | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HA-BSI: Patients with HA-BSI treated in an ICU
  Interventions: Other: Treatment

INTERVENTIONS:
Other: Treatment — Antimicrobial and other treatment modalities such as source control, vasoactive medications, dialysis

SUMMARY:
In this observational study, it is aimed to investigate the mortality and morbidity rates of hospital-acquired blood stream infections that are treated in intensive care units (ICU). The effects of properties of the micro-organism such as type and antimicrobial resistance on the infection and its outcomes will be mainly explored. In addition, the impact of antibiotic options and other treatment modalities on survival of patients will be investigated. Twenty-seven different ICUs from Turkey will be included in this study.

DETAILED DESCRIPTION:
Blood stream infection (BSI) is defined as the identification of a culprit pathogen in the blood culture sample of a participant. As such, and once contaminants are excluded, BSI is the only cause of sepsis where the presence of an infection and the pathogen are known with certainty. This makes BSI the perfect model of infection to study the effects of the micro-organism on the participant, and the effects of the antibiotics and other treatments on survival. There is an increasing trend in antimicrobial resistance rates among microorganisms that are associated with nosocomial infections treated in ICU. However, infectious diseases physicians from Turkey do not know contemporary epidemiological data of hospital-acquired BSI treated in ICU in Turkey.

This study 'Epidemiology and Determinants of Outcomes of Hospital-Acquired Blood Stream Infections in the Intensive Care in Turkey' is a multi-center prospective observational cohort study that will include patients with hospital-acquired blood stream infections (HA-BSI) treated in ICUs in Turkey. This study will present unknown current epidemiology of HA-BSI in Turkey. Furthermore, It will provide very important data about 28-day mortality rates of HA-BSI treated in ICU. The primary outcomes of this study can be accounted as following: (i)determinants of outcomes of HA-BSI, (ii) the effects of the source of infection on outcomes, (iii) the effects of microorganism on these outcomes, (iv) the effects of antimicrobial therapy and of source control on investigated outcomes. In this study, participant specific and organizational factors will be explored and the determinants of management of HA-BSI in ICUs will be described.

There will be no intervention in this study. The data of participants will be obtained from hospital database and recorded into electronic case report forms anonymously.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 Years.
* Hospital Acquired Bloodstream Infection (HA-BSI).
* Treated in the ICU.
* ICU acquired OR Hospital acquired prior to ICU admission

Exclusion Criteria:

* Patients that had a positive blood culture in the hospital and transferred to ICU for a different reason than specific treatment of the causes or consequences of HA-BSI.
* Previous inclusion in the study.
* HA-BSI is defined as a positive blood culture (BC) sampled after 48 hours following hospital admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a HA-BSI treated in an ICU
Sampling Method: Non-Probability Sample
Enrollment: 810 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Mortality Rate | 28-day mortality
  Rate of all cause mortality

SECONDARY OUTCOMES:
Progress of organ failures | 7-day
  Assessed by the components of the Sequential Organ Failure Assessment (SOFA) score, minimum (0 point)- Maximum (24 points)
Days free or organ supportive therapy | 28-day
  Days free of renal replacement therapy, mechanical ventilation, vasopressors, intensive care unit
Rate of Clinical cure | 7-day and 28-day
  As evaluated by the treating clinician. There will be no specific tool for evaluation of clinical cure. It will be only determined by the clinical assessment of admitting physicians.
Rate of Microbiological cure | 7-day and 28-day
  Presence of persisting or relapsing blood stream infection

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Vincent JL, Rello J, Marshall J, Silva E, Anzueto A, Martin CD, Moreno R, Lipman J, Gomersall C, Sakr Y, Reinhart K; EPIC II Group of Investigators. International study of the prevalence and outcomes of infection in intensive care units. JAMA. 2009 Dec 2;302(21):2323-9. doi: 10.1001/jama.2009.1754. PMID 19952319
- [Background] Tabah A, Koulenti D, Laupland K, Misset B, Valles J, Bruzzi de Carvalho F, Paiva JA, Cakar N, Ma X, Eggimann P, Antonelli M, Bonten MJ, Csomos A, Krueger WA, Mikstacki A, Lipman J, Depuydt P, Vesin A, Garrouste-Orgeas M, Zahar JR, Blot S, Carlet J, Brun-Buisson C, Martin C, Rello J, Dimopoulos G, Timsit JF. Characteristics and determinants of outcome of hospital-acquired bloodstream infections in intensive care units: the EUROBACT International Cohort Study. Intensive Care Med. 2012 Dec;38(12):1930-45. doi: 10.1007/s00134-012-2695-9. Epub 2012 Sep 26. PMID 23011531
- [Background] De Waele JJ, Akova M, Antonelli M, Canton R, Carlet J, De Backer D, Dimopoulos G, Garnacho-Montero J, Kesecioglu J, Lipman J, Mer M, Paiva JA, Poljak M, Roberts JA, Rodriguez Bano J, Timsit JF, Zahar JR, Bassetti M. Antimicrobial resistance and antibiotic stewardship programs in the ICU: insistence and persistence in the fight against resistance. A position statement from ESICM/ESCMID/WAAAR round table on multi-drug resistance. Intensive Care Med. 2018 Feb;44(2):189-196. doi: 10.1007/s00134-017-5036-1. Epub 2017 Dec 29. PMID 29288367
- [Background] PRISM Investigators; Rowan KM, Angus DC, Bailey M, Barnato AE, Bellomo R, Canter RR, Coats TJ, Delaney A, Gimbel E, Grieve RD, Harrison DA, Higgins AM, Howe B, Huang DT, Kellum JA, Mouncey PR, Music E, Peake SL, Pike F, Reade MC, Sadique MZ, Singer M, Yealy DM. Early, Goal-Directed Therapy for Septic Shock - A Patient-Level Meta-Analysis. N Engl J Med. 2017 Jun 8;376(23):2223-2234. doi: 10.1056/NEJMoa1701380. Epub 2017 Mar 21. PMID 28320242